CLINICAL TRIAL: NCT05326022
Title: Microcurrent Therapy Versus Low-Level Laser Therapy on Post-surgical Wound Healing
Brief Title: Microcurrent Therapy and Low-Level Laser Therapy on Wound Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nehad Ahmed Youness Abo-zaid (Other)
Responsible Party: Sponsor-Investigator, Nehad Ahmed Youness Abo-zaid, Assistant professor of physical therapy, South Valley University
Organization: South Valley University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002599
Record Dates: First submitted 2022-03-23; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Wound Healing Delayed
MeSH Terms: interventions — Low-Level Light Therapy; Nutrition Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- medical therapy group (Experimental): formed of 20 patients to whom ordinary medical therapy as the pervious groups and placebo shame laser had been applied.
  Interventions: Other: Medical therapy
- medical therapy and Microcurrent group (Experimental): formed of 20 patients to whom the microcurrent therapy had been applied with ordinary medical therapy.
  Interventions: Device: Microcurrent therapy; Other: Medical therapy
- medical therapy and Low-Level Laser Therapy group (Experimental): formed of 20 patients to whom the Low Level Laser Therapy had been applied with ordinary medical therapy.
  Interventions: Device: Low Level Laser Therapy; Other: Medical therapy

INTERVENTIONS:
Device: Microcurrent therapy — Microcurrent therapy
  Arms: medical therapy and Microcurrent group
Device: Low Level Laser Therapy — Laser therapy
  Arms: medical therapy and Low-Level Laser Therapy group
Other: Medical therapy — Medical therapy

SUMMARY:
The study aiming to compare between the Microcurrent and Low-Level Laser Therapy on wound healing

DETAILED DESCRIPTION:
The study designed to compare between the Microcurrent and Low-Level Laser Therapy on wound healing

ELIGIBILITY:
Inclusion Criteria:

* patient recently undergo appendectomy

Exclusion Criteria:

* patient with neurological disorders
* patient with metabolic disorders

Ages: 10 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-04-28 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
levels of matrix metalloproteinases | assessed at day 3 post operative
  analyze by Enzyme-linked immunosorbent assay

SECONDARY OUTCOMES:
levels of matrix metalloproteinases | assessed at day 30 post operative
  analyze by Enzyme-linked immunosorbent assay
the tissue inhibitors of metalloproteinases | assessed at day 3 post operative
  analyze by Enzyme-linked immunosorbent assay
the tissue inhibitors of metalloproteinases | assessed at day 30 post operative
  analyze by Enzyme-linked immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A. Abo-Zaid, PhD, Principal Investigator — South Valley University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dickinson LE, Gerecht S. Engineered Biopolymeric Scaffolds for Chronic Wound Healing. Front Physiol. 2016 Aug 5;7:341. doi: 10.3389/fphys.2016.00341. eCollection 2016. PMID 27547189